CLINICAL TRIAL: NCT02162043
Title: Development and Evaluation of a Self-administered/Assisted Visual Field Screening Tool for Glaucoma
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Emmanouil Tsamis, Research Assistant, University of Manchester
Other Study IDs: 2366
Record Dates: First submitted 2014-06-06; First posted 2014-06-12 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Glaucoma; Diagnostic Self-evaluation
Keywords: Glaucoma; Perimetry; Diagnostic self-evaluation; Screening; Visual fields
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Usability assessment: Patients without any experience with visual field testing will be recruited and tested with different versions of the developed self-test. This will help identify usability features that will make the test user-friendly.
- Hospital-based clinical trial: The new test will be evaluated on patients attending Manchester Royal Eye Hospital to provide an estimate of its diagnostic performance.
- Community-based trial: Patients attending Manchester Royal Eye Hospital's outpatient clinics will be recruited to trial the new test on their friends and family in order to evaluate the uptake and performance of the new test in a home environment without any researchers/clinicians presence.

SUMMARY:
This project aims to evaluate a self-administered screening test for glaucoma, the second largest cause of blindness in the western world. New approaches to glaucoma screening are needed because a significant number of patients first present to hospitals with advanced-stage glaucoma and late presentation is associated with a much higher risk for future blindness. This project will develop a new user-friendly visual field test that will be made available through the internet for self-testing. It will conduct both hospital-based and community-based clinical trials to establish benefits and costs of this new test.

DETAILED DESCRIPTION:
Objectives: At a recent (19/4/2013) Priority Setting Partnership workshop, facilitated by the James Lind Alliance, patients, carers and eye health professionals produced a list of the top ten priorities for glaucoma research (http://www.sightlosspsp.org.uk/). Number 4 on the list was: What can be done to improve early diagnosis of sight-threatening glaucoma? The overarching aim of this project is to develop and evaluate a new visual field screening self-test that can be used to improve the early detection of glaucoma and thereby meet one of the aims of the Priority Setting Partnership. We will conduct hospital- and community-based clinical trials on the new test to establish its performance.

Methodology: This project will clinically evaluate the new test deriving measures of sensitivity and specificity. These trials will be conducted on patients attending the outpatient department of Manchester Royal Eye Hospital (MREH) and will use simulated defects to link performance measure with the extent of field damage. Patients without any established field loss will be tested. On completion of hospital-based clinical trials we will undertake locally based community trials to establish performance when self-administered or administered with the aid of friends/family, i.e. without researcher/clinician involvement. We will make the test available (emailed attachment that will install the test on the patients PC, laptop, tablet) to patients attending the glaucoma clinics of MREH with a request to test their friends and relatives. Guidance notes will emphasise the increased risk of developing glaucoma in blood relatives and the increased risk with age to help them target those at higher risk of developing glaucoma. Those failing the screening test, twice, will then undergo further testing by one of the Glaucoma Referral Refinement optometrists in Manchester to derive estimates of true and false referral rates.

ELIGIBILITY:
For the usability trials:

Inclusion Criteria:

* No visual field defects
* No previous visual field testing

Exclusion Criteria:

* Visual field defects MD>2dB
* Previous visual field testing experience

For the hospital-based trials:

Inclusion Criteria:

* No visual field defects

Exclusion Criteria:

* Visual field defects MD>2dB

For the community-based trials:

Exclusion Criteria:

* Subject not owning a PC or tablet

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the usability trials, volunteers with no previous perimetric experience will be recruited. Subjects will be based at Greater Manchester area.
  For the hospital- and community- based trials subjects will be recruited by Manchester Royal Eye Hospital's outpatient clinic
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2014-11; Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of the new self-test for glaucoma screening. | Two years
  We will measure the diagnostic performance of the new test to a range of simulated defects. We will establish the take up rate and number of true and false positives of the community trial when promoted through patients attending the glaucoma clinics of MREH.

SECONDARY OUTCOMES:
Diagnostic performance of the new test on patients suspect to glaucoma | Two years
  Throughout the development of this screening test, the research will, also, question whether or not the software could be adapted for use on suspect patients currently seen within the Hospital Eye Services (HES).

CONTACTS AND LOCATIONS:
Overall Officials: Prof David B Henson, Study Director — University of Manchester; Emmanouil Tsamis, Principal Investigator — University of Manchester
Locations (1):
- Royal Eye Hospital, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No